CLINICAL TRIAL: NCT02291913
Title: Phase II Open Label Study of Everolimus in Combination With Anti-estrogen Therapy in Hormone Receptor-Positive HER2-Negative Advanced Breast Cancer
Brief Title: Everolimus Combined With Anti-estrogen Therapy in Hormone-Receptor-Positive HER-2 Negative Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 212
Record Dates: First submitted 2014-11-10; First posted 2014-11-17 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: ER-Positive Breast Cancer; HER2-Negative Breast Cancer; everolimus; anti-estrogen therapy; PR-Positive Breast Cancer; Afinitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane; Tamoxifen; Fulvestrant; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- everolimus (Experimental): Everolimus will be administered at a dose of 10 mg PO daily combined with any one of the following anti-estrogen therapies on which the patient most recently progressed (tamoxifen, fulvestrant, anastrozole, letrozole, exemestane, toremifine, or LHRH agonists in conjunction with anti-estrogen therapy). Anti-estrogen therapy will be administered at the US Food and Drug Administration (FDA) prescribed doses.
  Interventions: Drug: Everolimus; Drug: Exemestane; Drug: Tamoxifen; Drug: Fulvestrant; Drug: Anastrozole; Drug: Letrozole; Drug: Toremifine

INTERVENTIONS:
Drug: Everolimus
  Other Names: Afinitor
Drug: Exemestane — Anti-estrogen therapy
Drug: Tamoxifen — Anti-estrogen therapy
Drug: Fulvestrant — Anti-estrogen therapy
Drug: Anastrozole — Anti-estrogen therapy
Drug: Letrozole — Anti-estrogen therapy
Drug: Toremifine — Anti-estrogen therapy

SUMMARY:
Many patients with ER-positive or PR-positive breast cancer are treated with endocrine therapy. Although most ER/PR-positive tumors initially respond to hormonal therapy, patients often experience disease progression. Everolimus, in combination with exemestane, has shown activity in endocrine-resistant disease. This study will evaluate the efficacy of Everolimus+ anti-estrogen therapy in patients with ER-positive metastatic breast cancer who have progressed after receiving anti-estrogen therapy.

DETAILED DESCRIPTION:
This is a multi-centered, open-labeled, Phase II study on metastastic breast cancer (MBC). The patient population includes locally recurrent or MBC patients with cytologically or histologically confirmed hormone receptor-positive breast cancer who have demonstrated disease progression on prior anti-estrogen therapy or therapies. Investigators propose to evaluate the efficacy of Everolimus in patients with ER-positive (estrogen receptor-positive) metastatic breast cancer who have progressed on anti-estrogen therapy. Forty-six (46) patients are planned for enrollment in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of unresectable, locally recurrent or MBC.
2. ER and/or PR-positive tumors with staining by immunohistochemistry (IHC) based on the most recent biopsy.
3. Only 1 previous chemotherapy regimen for MBC. Patients progressing while receiving adjuvant endocrine therapy or progressing <12 months from completion of adjuvant endocrine therapy are eligible.
4. Progressed on anti-estrogen therapy (tamoxifen, fulvestrant, anastrozole, letrozole, exemestane, toremifine, or LHRH agonists in conjunction with anti-estrogen therapy) defined as:

   * Recurrence while on, or within 12 months of end of anti-estrogen therapy for early stage breast cancer, or
   * Progression while on, or within one month of anti-estrogen therapy for locally advanced or metastatic breast cancer.

   Note: No washout for anti-estrogen therapy required. Anti-estrogen therapy does not have to be the last treatment prior to study entry.
5. Post-menopausal or pre/peri-menopausal women on tamoxifen. LHRH agonists may be used to render ovarian suppression with postmenopausal ranges of estradiol or FSH per institutional guidelines.
6. HER2-negative breast cancer, defined as follows:

   * Fluorescent In Situ Hybridization (FISH)-negative (FISH ratio <2.0), or
   * IHC 0-1+, or
   * IHC 2-3+ AND FISH-negative (FISH ratio <2.0).
7. Measureable disease as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 or evaluable bone lesions, lytic or mixed, in absence of measureable disease by RECIST criteria.
8. Adequate hematologic, hepatic and renal function.
9. International normalized ratio (INR) ≤1.5 or prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits (WNL) of the institution (if patient is not on anti-coagulation therapy).
10. Age ≥ 18 years.
11. ECOG Performance Status score of 0-2.
12. Life expectancy of ≥ 12 weeks.

Exclusion Criteria:

1. Previous therapy or known intolerance/hypersensitivity with any approved or investigational mTOR inhibitor (e.g., temsirolimus, everolimus, sirolimus).
2. Patients who are ≤21 days after their most recent chemotherapy and have not recovered from side effects.
3. Use of an investigational drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of everolimus. For investigational drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the investigational drug and administration of everolimus is required.
4. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days for metastatic disease prior to first dose of everolimus or has not recovered from side effects of such therapy.
5. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if there is no evidence of central nervous system (CNS) disease progression, and at least 2 weeks have elapsed since treatment. Patients are not permitted to receive enzyme inducing anti-epileptic drugs (EIAEDs) during the study and should not be receiving chronic corticosteroid therapy for CNS metastases.
6. Patients with known active hepatitis B (HBV) or hepatitis C (HCV) infection. Patients with risk factors for hepatitis must have HBV DNA and HCV RNA testing by PCR, and are ineligible if these tests are positive.
7. Patients receiving immunization with attenuated live vaccines within 1 week of study entry or during study period.

NOTE: There are additional inclusion/exclusion criteria. The study center will determine patient eligibility and respond to any questions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Study Chair — SCRI Development Innovations, LLC
Locations (8):
- United States (8):
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Memorial Cancer Center, Hollywood, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists-East, West Palm Beach, Florida
  - Hope Cancer Center, Terre Haute, Indiana
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2014 to December 2015, 48 patients who had locally recurrent or metastatic breast cancer with cytologically or histologically confirmed hormone receptor-positive breast cancer who have demonstrated disease progression on prior anti-estrogen therapy. Study was closed after enrollment goal was reached.
Groups:
- Everolimus: Everolimus will be administered at a dose of 10 mg PO daily combined with any one of the following anti-estrogen therapies on which the patient most recently progressed (tamoxifen, fulvestrant, anastrozole, letrozole, exemestane, toremifine, or LHRH agonists in conjunction with anti-estrogen therapy). Anti-estrogen therapy will be administered at the US Food and Drug Administration (FDA) prescribed doses.
  Everolimus
  Exemestane: Anti-estrogen therapy
  Tamoxifen: Anti-estrogen therapy
  Fulvestrant: Anti-estrogen therapy
  Anastrozole: Anti-estrogen therapy
  Letrozole: Anti-estrogen therapy
  Toremifine: Anti-estrogen therapy
Period: Overall Study
Arm/Group | Everolimus
Started | 48
Completed | 0
Not Completed | 48
Not completed — Progressive Disease | 32
Not completed — Adverse Event | 11
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of treatment.
Groups:
- Everolimus: Everolimus will be administered at a dose of 10 mg by mouth daily combined with any one of the following anti-estrogen therapies on which the patient most recently progressed (tamoxifen, fulvestrant, anastrozole, letrozole, exemestane, toremifine, or LHRH agonists in conjunction with anti-estrogen therapy). Anti-estrogen therapy will be administered at the US Food and Drug Administration (FDA) prescribed doses. A treatment cycle was defined as 4 weeks, with radiological evaluations every 8 weeks.
  Everolimus
  Exemestane: Anti-estrogen therapy
  Tamoxifen: Anti-estrogen therapy
  Fulvestrant: Anti-estrogen therapy
  Anastrozole: Anti-estrogen therapy
  Letrozole: Anti-estrogen therapy
  Toremifine: Anti-estrogen therapy
Arm/Group | Everolimus
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the time from Day 1 of study drug administration to disease progression as defined by RECIST (Response Evaluation Criteria in Solid Tumors) version 1.1 criteria, or death on study. Participants who are alive and free from disease progression will be censored at the date of last radiologic tumor assessment. Participants who receive non-protocol therapy (subsequent therapy) prior to incurring an event will be censored at the date of last tumor assessment prior to the start of subsequent therapy. Participants who do not have a post-baseline tumor assessment will be censored at the date of first treatment (Day 1).
Time Frame: up to 3 years
Population: Participants who received at least 1 cycle of study treatment and had at least one post-baseline radiologic assessment were evaluable for PFS analysis per protocol. 36 of the total 48 patients were analyzed for PFS. The remaining 12 treated patients did not meet this criteria to be analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 36
months | 7.2 [4.1 to 10.0]

2. Secondary Outcome: Number of Patients With Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: Assessments were made through analysis of the reported incidence of treatment-emergent AEs. All participants who received at least one dose of protocol treatment were followed for safety. Adverse events were collected from day of first dose to 30 days after last protocol treatment and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Up to 20 months
Population: Number of participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 48
Participants | 48

3. Secondary Outcome: Number of Patients With an Objective Response (CR or PR) Also Called the Overall Response Rate (ORR).
Description: Defined as the number of patients with objective evidence of complete or partial response (CR or PR) using RECIST version 1.1. A CR is the complete disappearance of all target lesions. A PR is a decrease of 30% or more of the diameter(s) of all target lesions from the baseline sum of diameters.
Time Frame: every 8 weeks until discontinuation, up to 20 months
Population: Participants who received at least 1 cycle of study treatment and had at least one post-baseline radiologic assessment. 36 of the total 48 patients were analyzed for PFS. The remaining 12 treated patients did not meet this criteria to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 36
Participants | 2

4. Secondary Outcome: Number of Participants With CR, PR, or 6 Months of SD Also Called Clinical Benefit Rate (CBR)
Description: The proportion of patients with Complete Response (CR) or Partial Response (PR) or 6 months or more of Stable Disease (SD). A CR is the complete disappearance of all target lesions. A PR is a decrease of 30% or more of the diameter(s) of all target lesions from the baseline sum of diameters. SD is not meeting the criteria for PR or a 20% increase in target lesions called Progressive Disease (PD).
Time Frame: Up to 20 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 36
Participants | 12

5. Secondary Outcome: Median Time From First Occurrence of CR or PR to Disease Progression or Death Also Called Duration of Response (DOR)
Description: Only those patients who achieved Complete Response or Partial Response will be included in the summaries of DOR. DOR is defined as time from first date of response of CR or PR to disease progression or death as defined by RECIST v1.1 criteria. Participants who are alive and free from disease progression will be censored at the date of last tumor assessment. Patients who receive non-protocol therapy (subsequent therapy) prior to incurring an event will be censored at the date of last tumor assessment prior to the start of subsequent therapy. A CR is the complete disappearance of all target lesions. A PR is a decrease of 30% or more of the diameter(s) of all target lesions from the baseline sum of diameters.
Time Frame: every 8 weeks until discontinuation, up to 20 months
Population: Only those patients who achieved Complete Response or Partial Response will be included in the summaries of DOR. A CR is the complete disappearance of all target lesions. A PR is a decrease of 30% or more of the diameter(s) of all target lesions from the baseline sum of diameters.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 2
months | 8.8 [1.8 to 11.8]

6. Secondary Outcome: Median Overall Survival (OS)
Description: Defined as the time from date of first study treatment to date of death due to any cause. Patients who are alive will be censored at the date of last known date alive.
Time Frame: up to 3 years from first treatment
Population: Participants who received at least 1 cycle of study treatment and had at least one post-baseline radiologic assessment were evaluable for OS analysis per protocol. 36 of the total 48 patients were analyzed for OS. The remaining 12 treated patients did not meet this criteria to be analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 36
months | 26.7 [16.3 to 26.7]

ADVERSE EVENTS:
Time Frame: Up to 20 months
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from day of first dose to 30 days after last protocol treatment and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 32/48
Serious Adverse Events (participants affected / at risk) | 15/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=48)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Non-Cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=48)
Fatigue (General disorders) | 31
Nausea (Gastrointestinal disorders) | 18
Stomatitis (Gastrointestinal disorders) | 15
Rash (Skin and subcutaneous tissue disorders) | 15
Mucosal Inflammation (General disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 12
Headache (Nervous system disorders) | 11
Vomiting (Gastrointestinal disorders) | 10
Urinary Tract Infection (Infections and infestations) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Anaemia (Blood and lymphatic system disorders) | 8
Decreased Appetite (Metabolism and nutrition disorders) | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7
Insomnia (Psychiatric disorders) | 7
Oedema Peripheral (General disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Aspartate Aminotransferase Increased (Investigations) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 3
Cellulitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Alanine Aminotransferase Increased (Investigations) | 3
Weight Decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Depression (Psychiatric disorders) | 3
Rash Pruritic (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2014-06-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT02291913/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT02291913/SAP_001.pdf